CLINICAL TRIAL: NCT01155180
Title: Leptin in the Maintenance of Reduced Body Weight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Christos Mantzoros, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008P000190; R01DK079929 (NIH)
Record Dates: First submitted 2010-06-16; First posted 2010-07-01 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Leptin; metreleptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leptin (Experimental): We will start the leptin at a dose of 0.08mg/kg fat mass in men and 0.14mg/kg fat mass in women
  Interventions: Drug: Leptin
- Placebo (Placebo Comparator): We will start the placebo at a dose of 0.08mg/kg fat mass in men and 0.14mg/kg fat mass in women
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Leptin — Hormone - daily self injections for 6 months
  Other Names: metreleptin
  Arms: Leptin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
You are invited to take part in a research study about the role of leptin (a fat cell hormone that normally circulates in the blood) on maintaining a reduced body weight. This study will also evaluate how leptin impacts hormone levels, metabolic rate (how many calories are used at rest), autonomic nervous function (the part of your brain that controls your heart rate and breathing), changes in body composition and your sense of appetite. Under normal conditions, leptin is secreted by fat cells and signals to the brain to decrease appetite and regulate energy usage and hormone levels. When obese individuals lose weight, their leptin levels go down, which may cause them to later regain the weight. This study will provide leptin as an investigational medication (not yet approved by the Food and Drug Administration) to increase the levels of the leptin hormone that normally circulates in your blood back to a normal range. We will see if this can help you to maintain your reduced body weight and improve your hormonal and metabolic function.

DETAILED DESCRIPTION:
Study Overview This study is a randomized, double-blind, placebo-controlled study of leptin administration to individuals with a recent 10% weight loss, achieved through lifestyle intervention program. In this study proposal, we propose that 90 subjects who have recently completed a lifestyle intervention weight loss program (at one of the four participating Boston Weight loss centers) and have achieved a weight loss of more than 10% body weight will be enrolled in the study. They will have baseline studies performed (including full neuroendocrine evaluation as described below) and will be randomized to leptin/placebo in the ratio 1:1 after stratification by center. They will continue to receive standard weight maintenance advice with intermittent nutrition and behavioral counseling. Our aim is to finally study a total of 36 subjects per treatment arm (20% drop out or inability to achieve and/or maintain10% weight loss expected). Leptin levels will be checked every month and the dose will be titrated to achieve and keep serum levels equivalent to those at baseline based on baseline weight. We will start the leptin/placebo at a dose of 0.08mg/kg fat mass in men and 0.14mg/kg fat mass in women, with dose titration to achieve baseline leptin levels utilizing formulas derived from our pharmacokinetic studies Leptin levels will be checked every month. Circulating leptin levels between +30% and -10% of baseline will be considered acceptable. Otherwise, the leptin dose will be adjusted accordingly. Our aim is to keep the mean leptin level at or within +30% of baseline. Subjects will be studied prior to receiving leptin, after four weeks and six months of weight maintenance and we will compare changes in body weight and composition, neuroendocrine function, and metabolic function between the leptin and placebo-treated groups. In addition, the first 23 subjects per group will have measurement of total energy expenditure performed using doubly labeled water at baseline and 6 months. This will allow us to examine the effects of leptin replacement, to levels observed at baseline body weight, on the maintenance of weight loss and the neuroendocrine and metabolic adaptation to decreasing body weight in obese individuals. While difference in weight maintenance at six months will be our primary outcome, subjects will also be studied after 4 weeks of weight maintenance, which will allow us to determine the role of leptin in the adaptation to weight loss under stable, weight maintenance conditions. We have chosen the four week time point as previous nonrandomized, uncontrolled studies have been able to document an effect of leptin replacement after this time. Both groups will be followed for an extended 6-month period during which they will receive standard weight maintenance advice, in addition to leptin/placebo. We will observe the changes in weight, neuroendocrine function, metabolic function and leptin signaling over this time and compare the leptin and placebo groups. In this subset of 23 subjects per group we will evaluate energy expenditure by doubly labeled water. Finally, subjects will be followed for a further 6 months after the end of the study to document further changes in body weight as an additional study outcome.

ELIGIBILITY:
Inclusion criteria for dietary induced weight loss group:

* Age 18 or older
* Body mass index (pre weight loss) between 30 and 40 kg/m2.
* Weight loss achieved over a period not greater than 6 months.

Exclusion criteria for dietary induced weight loss group:

* Use of a very low calorie diet in the year prior to the start of the study
* History of diabetes
* History of any illness that may affect the concentrations of the hormones to be studied (such as anemia, infectious diseases, renal or hepatic failure, cancer, lymphoma, clinically evident hypogonadism, malabsorption or malnourishment, hypo or hyperthyroidism, hypercortisolism, alcoholism or drug abuse, eating disorders)
* On medications known to affect the hormones to be measured in this study (such as glucocorticoids, anti seizure medications or thyroid hormones), or medications for weight loss.
* Known history of reactions or known hypersensitivity to E. Coli derived proteins
* Breast feeding, pregnant, or wanting to become pregnant during the next year
* Subjects with any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g. cochlear implants, pacemakers, neuron or biostimulators, electronic infusion pumps, etc.).
* Subjects with any type of ferromagnetic bioimplant that could potentially be displaced or damaged, such as aneurysm clips, metallic skull plates, etc.
* Subjects that exhibit noticeable anxiety and/or claustrophobia.
* Subjects who have cardiac or known circulatory impairment, and/or the inability to perspire (poor thermoregulatory function).
* Subjects who have significant sensory or motor impairment; - Subjects who suffer from epilepsy, in particular photo-sensitive epilepsy (this would be a risk for scanning with visual stimulation).
* Subjects with neurological problems that might interfere or complicate testing (e.g. presence of titubation).
* Subjects who cannot adhere to the experimental protocol for any reason.

Inclusion criteria for lap band surgery induced weight loss group:

* Age 18 or older.
* Body mass index (pre weight loss) between 30 and 40 kg/m2.
* Weight loss achieved over a period not greater than 6 months.
* Approved for bariatric surgery as per Beth Israel Deaconess Medical Center (BIDMC) Bariatric Clinic guidelines
* Adult men and women, age 18-65
* English speaking
* Willing and able to take part in a multi year study involving visits and telephone interviews
* Enrolled prior to bariatric surgery.

Exclusion Criteria:

* Any condition that would exclude a patient from lap band surgery as listed below -
* patients with untreated major depression or psychosis
* binge eating disorders
* current drug and alcohol abuse
* severe cardiac disease with prohibitive anesthetic risks
* severe coagulopathy i
* inability to comply with nutritional requirements including life-long vitamin replacement.
* pregnancy
* Any additional condition which is not in accordance with standard of care as per Bariatric Clinic at BIDMC.
* Any condition which in the opinion of the investigators makes the candidate unsuitable for participation in this study
* Diabetes controlled by medication

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos S Mantzoros, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who have successfully completed 1of the 4 hospital-based participating weight loss programs (Boston Medical Center, Tufts Medical Center, Massachusetts General Hospital, Beth Israel Deaconess Medical Center (BIDMC)-Joslin Center) & have achieved a >8% (average 10%, range 8-14%) weight loss will be invited to participate in the study.
Period: Overall Study
Arm/Group | Leptin | Placebo
Started | 18 | 6
Completed | 18 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: We will start the placebo at a dose of 0.08mg/kg fat mass in men and 0.14mg/kg fat mass in women
  Placebo: Placebo-daily self injections for 6 months
- Total: Total of all reporting groups
Arm/Group | Leptin | Placebo | Total
Number analyzed (Participants) | 18 | 6 | 24
Age, Customized [Mean (Full Range); unit: years]
  years | 32 [23 to 41] | 45.5 [24 to 67] | 45 [23 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 9 | 0 | 9
Region of Enrollment [Number; unit: participants]
  United States | 18 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight at 6 Months
Description: Body weight was recorded to the nearest 0.1 kg at baseline and at 6 months after randomization. Then the percentage change was calculated.
Time Frame: baseline and 6 months after randomization
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Leptin | Placebo
Number analyzed (Participants) | 18 | 6
percentage change | 10.2 (1.7) | 12.7 (1.2)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Leptin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6
Other Adverse Events (participants affected / at risk) | 0/18 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No